CLINICAL TRIAL: NCT00290082
Title: Comparison Between Midazolam and Loxapine in the Treatment of Agitated Patients in the Emergency Department
Brief Title: Randomized Double-blind Trial of Midazolam and Loxapine in Agitated Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: 2 complications with midazolam
Sponsor: University Hospital, Rouen (Other)
Responsible Party: CHU-Hopitaux de Rouen, Delegation de la recherche clinique
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004/055/HP; French state grant
Record Dates: First submitted 2006-02-09; First posted 2006-02-10 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Acute Agitated Patients
Keywords: sedation; midazolam; loxapine; agitation; emergency department; toxicological analysis
MeSH Terms: conditions — Psychomotor Agitation; Emergencies | interventions — Loxapine; Midazolam; Blood Specimen Collection; Remote Patient Monitoring

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- loxapine (Active Comparator): agitated patients were randomly assigned either to loxapine, either to midazolam group
  Interventions: Drug: loxapine, midazolam; Biological: blood sample; Other: patient monitoring; Drug: Loxapine
- midazolam (Active Comparator): midazolam is compared to loxapine in terms of efficacy and tolerance
  Interventions: Drug: loxapine, midazolam; Biological: blood sample; Other: patient monitoring; Drug: Midazolam

INTERVENTIONS:
Drug: loxapine, midazolam — agitated patients received loxapine 1 ml/ kg body weight ( loxapine 25mg/ml) or midazolam 1 ml/ kg body weight ( midazolam 1mg/ml) if patients were still agitated 20 min after the first treatment, they received loxapine 0.5 ml/ kg body weight ( loxapine 25mg/ml) or midazolam 0.5 ml/ kg body weight ( midazolam 1mg/ml)
  Other Names: Loxapac; Hypnovel
Biological: blood sample — was evaluated in patients sedated, alcohol level, blood sugar
  Other Names: Loxapac; Hypnovel
Other: patient monitoring — Till his coming out the emergency service, patient had an hemodynamic, respiratory and neurologic monitoring as well as an agitated score monitoring The occurence of a complication during the 15 days after leaving the emergency department was prospected.
Drug: Loxapine — Loxapine 1 mL / 10 kg
  Arms: loxapine
Drug: Midazolam — Midazolam 1 mL / 10 Kg
  Arms: midazolam

SUMMARY:
Neuroleptics are used since a long time in the management of severely agitated patients. Loxapine is routinely used in our country, with, to our knowledge no severe adverse event reported, in this indication.

However, recently, benzodiazepines have appeared interesting in agitated patients, with the use of midazolam.

The aim of this study is to compare midazolam to loxapine in the treatment of severe agitated patients admitted in the emergency department.

DETAILED DESCRIPTION:
Prospective, Randomized, Double-blind, Multicenter study (20 french emergency departments)

ELIGIBILITY:
Inclusion Criteria:

Severely agitated patients (Richard Scale over or equal to 5) between 18 and 65 years old

Exclusion Criteria:

Hypoglycemia hypoxemia patients with known dementia blood pressure <90 mmHg known cocaine or amphetamine intoxication pregnancy respiratory or liver insufficiency myasthenia sedation before arrival to hospital

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Success of treatment at 20 min | 20 min

SECONDARY OUTCOMES:
Success of treatment at 40 and 60 min | 40 and 60 mn
Agitation level at 20,40 and 60 min | 20, 40 and 60mn
Need for rescue medication | any time
Sedation duration
treatment failure | one hour after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fabienne FM Moritz, MD, Principal Investigator — University Hospital, Rouen
Locations (21):
- France (21):
  - Emergency Department, Créteil, Paris
  - Emergency Department, Ghps, Paris
  - Emergency Department, Agen
  - Emergecy department, Argenteuil
  - Emergency Department, Bayeux
  - Emergency Department, Bondy
  - Emergency Department, Carcassonne
  - Emergency Department, Clermont-Ferrand
  - Emergency Department, Dijon
  - Emergency Department, Elbeuf
  - Emergency Department, Grenoble
  - Emergency Department, Le Havre
  - Emergency Department, Le Kremlin-Bicêtre
  - Emergency Department, Le Mans
  - Emergency Department, Lisieux
  - Emergency Department, Montauban
  - Emergency Department, Nantes
  - Emergency Department, Pontoise
  - Emergency Department, Raincy-Montfermeil
  - Emergency Department, Roanne
  - Emergency Department, Saint-Etienne